CLINICAL TRIAL: NCT05196178
Title: Effects of Spinal Cord Stimulation Therapy on Motor Function and Gait in Patients With Pure Hereditary Spastic Paraplegias
Brief Title: Spinal Cord Stimulation Therapy for Hereditary Spastic Paraplegias Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20211116
Record Dates: First submitted 2021-12-02; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-11

CONDITIONS: Motor Function; Gait
Keywords: spinal cord stimulation; Hereditary Spastic Paraplegias; Spasticity; gait
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Muscle Spasticity | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Spinal cord stimulation therapy (Experimental): Spinal cord stimulation at the thoracic levels ranging from T10 to T12.
  Interventions: Procedure: Spinal cord stimulation

INTERVENTIONS:
Procedure: Spinal cord stimulation — Paddle-shaped Spinal cord stimulation electrode with 16 contacts (AdaptiveStim® 39, 565;Medtronic, USA) will be implanted into the epidural space at the thoracic levels ranging from T10 to T12.

SUMMARY:
It's a single-center, prospective, open label clinical study with a 12 months follow-up period, to investigate the therapeutic effect and safety of spinal cord stimulation (SCS) on motor function and gait in patients with pure Hereditary Spastic Paraplegias.

DETAILED DESCRIPTION:
Pure hereditary spastic paraplegia is a heterogeneous group of genetic disorders characterized by degeneration of the corticospinal tracts, coursing with progressive weakness and spasticity of the lower limbs. The available anti spastic agents and surgical procedures involving anti-spastic systemic drugs, botulinum toxin, intrathecal baclofen, and even selective dorsal rhizotomy have not shown an improvement in muscle strength. Physical rehabilitation alone has shown positive results in short term, but this effect tends to fade away in few months.To date, there are no effective treatments for progressive deficits or disease-modifying therapy for Hereditary spastic paraplegia patients,

Spinal cord stimulation is a wellestablished therapy for the treatment of chronic neuropathic pain. Recently, some pilot studies demonstrated encouraging results of SCS in improving motor function. Patients severely affected by spinal cord injury experienced enhancements in leg movements and Parkinson's disease, primary progressive freezing of gait, and multiple system atrophy with predominant parkinsonism patients improved gait performance and freezing of gait after spinal cord stimulation by inducing changes in spinal and brain circuitry function. Some case studies suggest spinal cord stimulation may delay motor worsening and be innovative lines of research for the treatment of spastic paraplegia. However, evidence from larger numbers of subjects is still lacking. The objective of this study is to investigate the therapeutic effect and safety of spinal cord stimulation on motor function and gait in patients with pure hereditary spastic paraplegias

It's a single-center, prospective, open label clinical study with a 12 months follow- up period. The intended study population is individuals suffering from pure hereditary spastic paraplegia.Each participant will complete an enrollment/ screening/baseline visit, a spinal cord stimulation implant and activation visit, and a minimum of two follow-up visits, including visit at 3 months and the final study visit at 12months. The participants will proceed to implantation after satisfying implant inclusion and exclusion criteria. Paddle-shaped Spinal cord stimulation electrode with 16 contacts ((AdaptiveStim 39, 565; Medtronic, Minneapolis, USA) will be implanted into the epidural space at the thoracic levels ranging from T10 to T12. Electrode position will be verified by X-ray. The stimulators will be turned on within 1 month after electrode implantation surgery (slightly below sensory threshold). The stimulation parameters could vary freely, but medications will be kept constant during the study period. At the end of month 12, participants will enter the long-term follow-up in which medications and stimulation parameters could vary freely.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 14 and 70 years
2. patients with pure hereditary spastic paraplegias
3. with progressive weakness and spasticity of the lower limbs, and the gait dysfunction treatable by medication but not adequately controlled with medications
4. Understand potential risk/benefit, consent to the study, study procedures, and agree to complete the study follow-up visits and comply with the study protocol requirements.

Exclusion Criteria:

1. cognitive impairment ( MMSE≤24), depression (HAMD>24),acute psychosis, active alcohol or drug abuse, terminal illness, and any major medical or psychological histories, diagnoses, conditions, or comorbidities that would interfere with participation in the study per the investigatior's medical judgment
2. surgical or medical contraindications to spinal cord stimulation surgery(e.g. uncontrolled hypertension, advanced coronary artery disease).

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
change in spastic paraplegia rating scale(SPRS) | twelve months after surgery
  demonstrate the statistically significant improvement in score of spastic paraplegia rating scale(SPRS) from baseline( Off medication) to 12 months(On stimulation/Off medication); The score of SPRS ranges from 0 to 52, higher scores mean a worse outcome .

SECONDARY OUTCOMES:
change in the score of Modified Ashworth Scale | twelve months after surgery
  demonstrate statistically significant improvement in score of Modified Ashworth Scale from baseline( Off medication) to 12 months(On stimulation/Off medication); The score of Modified Ashworth Scale ranges from 0 to 4, higher scores mean a worse outcome.
change in Activities of Daily Living Scale (ADL) | twelve months after surgery
  demonstrate statistically significant improvement in score of Activities of Daily Living Scale (ADL) from baseline to 12 months. The score of ADL ranges from 0 to 100, higher scores mean a better outcome.
change in Tinetti Balance and Gait Analysis | twelve months after surgery
  demonstrate statistically significant improvement in the score of Tinetti balance and gait analysis from baseline( Off medication) to 12 months(On stimulation/Off medication); The score of Tinetti balance and gait ranges from 0 to 28, higher scores mean a better outcome.
change in Berg Balance Scale(BBS) | twelve months after surgery
  demonstrate statistically significant improvement in score of Berg Balance Scale(BBS) from baseline( Off medication) to On stimulation/Off medication state at 12 months. BBS ranged from 0 to 56, higher scores mean a better outcome.
Clinical Global Impression-Global Improvement | twelve months after surgery
  Evaluations will performed in off-stimulation and in on-stimulation conditions at 12 months after surgery on the basis of the physician's assessment, as well as on the basis of the patients'selfreported satisfaction. It is rated on a 7-point scale, range from 1(very much improved) through to 7 (very much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Zhang, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No